CLINICAL TRIAL: NCT02144168
Title: The Effect of Enteral Nutrition Supplemented With Prebiotics on Colonic Microbiota in the Critically Ill Patients: A Randomized Controlled Trial
Brief Title: The Effect of Enteral Nutrition Supplemented With Prebiotics on Colonic Microbiota in the Critically Ill Patients
Acronym: PrebioticFOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Mazuin Kamarul Zaman, Mrs, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PG127-2013A
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Diarrhoea
Keywords: Prebiotics; diarrhoea; Enteral nutrition; Fibre; Bifidobacteria; SCFA
MeSH Terms: conditions — Diarrhea | interventions — Osmolite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- prebiotics-free enteral formula (Active Comparator): Patients in this arm will be receiving standard, prebiotics-free enteral formula : Osmolite 1 cal
  Interventions: Dietary Supplement: Prebiotics-free enteral formula
- prebiotics containing enteral formula (Experimental): Patients in this arm will be receiving prebiotics containing enteral formula:Ensure Fos for 14 days
  Interventions: Dietary Supplement: Prebiotics containing enteral formula

INTERVENTIONS:
Dietary Supplement: Prebiotics-free enteral formula — Patient will be given Osmolite 1 cal for 2 weeks after baseline stool sample obtained
  Other Names: Osmolite 1 cal
  Arms: prebiotics-free enteral formula
Dietary Supplement: Prebiotics containing enteral formula — Patient will be given Ensure Fos for 2 weeks after baseline stool sample obtained
  Other Names: Ensure Fos
  Arms: prebiotics containing enteral formula

SUMMARY:
Primary objective of this study is to measure the change of concentration of faecal bifidobacteria between critically ill patients who receive enteral formula with and without prebiotics during enteral nutrition.Our null hypothesis is that there is no difference in the concentration of faecal bifidobacteria between critically ill patients who receive enteral formula with and without prebiotics during enteral nutrition (EN). Three faecal samples will be taken from the patient. First faecal sample is the first stool after initiation of EN and second sample is taken seven days after the initial sample and the third faecal sample is taken at day 14 after initial sample. Patient will be randomized to receive either of described formula after baseline (first) stool sample is obtained. Patient will be monitored up to 14 days after the initial stool sample is obtained.

DETAILED DESCRIPTION:
Written approval of the study has been obtained from the University Malaya Medical Centre (UMMC) Ethics Committee before commencement of this study

Patients will be screened for inclusion and exclusion criteria of the study and consent will be obtained from the patients or their legal representative in view of most critically ill patients are unconscious. Patients or their legal representative will be briefed regarding the objectives and the design of the study.

Critically ill patients recruited for this study will be exclusively on EN as clinically indicated. The volume of formula prescribed is based on each patient's total energy expenditure, which will be calculated by clinical dietitians. Formula will be delivered through a Ryles tube according to dietitians' order.

A faecal sample from the recruited patients will be collected for analysis at baseline, the first stool output after initiation of EN. Once baseline sample is collected, patients will be randomly assigned to receive enteral formula with or without prebiotics. Randomisation will be generated by using the website Randomization.com (http://www.randomization.com). Patients will be monitored for at least 14 days from passage of the first faecal sample after initiation of EN.

A faecal sample will be collected for analysis on days 0, 7, and 14. If there is absence of habitual or meal cues to stool output, samples will be collected and analyzed from each patient during 3 days periods at Day 6-8 for second faecal sample and Day 12-14 for the third faecal sample.

To guarantee accurate measurement of microbiota and shirt chain fatty acids (SCFA), only fresh faecal samples will be analyzed.Faecal samples will be collected within 1 hour of voiding and will immediately be transported to the laboratory for analysis of microbiota. The faecal sample will be homogenized using a sterile stainless steel Waring blender and aliquots of each specimen and will be frozen at -80°C until DNA is extracted.

Although the study is an open-label study, the researcher will be blinded for the analysis of the faecal sample for the quantification of faecal microbiota and short SCFA. An external Predominant component of the faecal microbiota; Bacteroides, Bifidobacteria, Clostridia and Lactobacilli will be quantified using Real Time Polymerase Chain Reaction (PCR). Faecal SCFA will be analyzed using gas-liquid chromatography, and C.difficile-enterotoxins A and B will be measured using enzyme-linked immunosorbent assay kit.

Faecal output will be recorded by nursing staff using a stool chart validated for use in this patient group. The chart will aid in the characterization of faecal frequency, consistency, and weight, which are then summarized into a daily stool score. A score of 15 or more is used to indicate diarrhoea (Whelan, Judd, Preedy, & Taylor, 2008). Patients will be visited once, daily during weekdays and contacted by telephone during weekends to monitor data recording by the nursing staff.

Details of EN regimen; formula used, amount, frequency, route and mode of delivery will be recorded progressively. Demographic data such as age sex, race and clinical details such as antibiotic, medications prescription and patients' progression will be extracted from the patients' medical notes daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving exclusive EN , nasogastric, continuous infusion
* Adult patients , 18 years old and above
* Critically ill patients
* Expected to require EN more than five days(Bleichner et al., 1997)

Exclusion Criteria:

* Patients with gastrointestinal disease (Sokol et al., 2006) or GIT surgery
* Patients receiving lactulose (Bouhnik et al., 2004)
* Currently under chemotherapy treatment (Kapkac et al., 2003)
* Patients who had received prebiotics and probiotics supplements within the previous one month
* Patients who have diarrhoea, 3 consecutive days (Majid et al, 2013)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of diarrhoea | up to 14 days post intervention

SECONDARY OUTCOMES:
Changes in faecal microbiota | baseline, 1 week & 2 weeks after baseline sample

OTHER OUTCOMES:
Changes in short chain fatty acid | baseline, 1 week & 2 weeks after baseline sample

CONTACTS AND LOCATIONS:
Overall Officials: Mazuin Kamarul Zaman, BSc (RD), Principal Investigator — University of Malaya; Hazreen Abdul Majid, BSc(RD),PhD, Principal Investigator — University of Malaya; Vineya Rai Hakumat Rai, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Petaling Jaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Bleichner G, Blehaut H, Mentec H, Moyse D. Saccharomyces boulardii prevents diarrhea in critically ill tube-fed patients. A multicenter, randomized, double-blind placebo-controlled trial. Intensive Care Med. 1997 May;23(5):517-23. doi: 10.1007/s001340050367. PMID 9201523
- [Background] Sokol H, Seksik P, Rigottier-Gois L, Lay C, Lepage P, Podglajen I, Marteau P, Dore J. Specificities of the fecal microbiota in inflammatory bowel disease. Inflamm Bowel Dis. 2006 Feb;12(2):106-11. doi: 10.1097/01.MIB.0000200323.38139.c6. PMID 16432374
- [Background] Bouhnik Y, Attar A, Joly FA, Riottot M, Dyard F, Flourie B. Lactulose ingestion increases faecal bifidobacterial counts: a randomised double-blind study in healthy humans. Eur J Clin Nutr. 2004 Mar;58(3):462-6. doi: 10.1038/sj.ejcn.1601829. PMID 14985684
- [Background] Kapkac, M., Erikoglu, M., Tuncyurek, P., Ersin, S., Esassolak, M., Alkanat, M., & Sipahioglu, O. (2003). Fiber enriched diets and radiation induced injury of the gut. Nutrition research (New York, N.Y.), 23(1), 77-83
- [Background] Whelan K, Judd PA, Preedy VR, Taylor MA. Covert assessment of concurrent and construct validity of a chart to characterize fecal output and diarrhea in patients receiving enteral nutrition. JPEN J Parenter Enteral Nutr. 2008 Mar-Apr;32(2):160-8. doi: 10.1177/0148607108314769. PMID 18407909
- [Background] Majid HA, Cole J, Emery PW, Whelan K. Additional oligofructose/inulin does not increase faecal bifidobacteria in critically ill patients receiving enteral nutrition: a randomised controlled trial. Clin Nutr. 2014 Dec;33(6):966-72. doi: 10.1016/j.clnu.2013.11.008. Epub 2013 Nov 16. PMID 24290345